CLINICAL TRIAL: NCT06661967
Title: Topical Oral Anesthesia Adjuncts in Conventional Intubation: A Randomized Controlled Trial Evaluating the Impact of Topical Oral Anesthesia on First-pass Success Rate
Brief Title: Topical Oral Anesthesia Adjuncts in Conventional Intubation on First-Pass Success Rate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 017/2567
Record Dates: First submitted 2024-10-23; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Unrecognized Condition

STUDY DESIGN:
Intervention Model Description: The participants are randomized into two groups. The first group receives lidocaine oral spray during preoxygenation while the latter will receive NSS spray as placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine spray (Active Comparator): Spray lidocaine 10 puffs at oropharynx during preoxygenation if the patient body weight is lower than 60kg, otherwise 15 puffs
  Interventions: Drug: Lidocaine spray
- Placebo (Placebo Comparator): Spray normal saline 10 puffs at oropharynx during preoxygenation if the patient body weight is lower than 60kg, otherwise 15 puffs
  Interventions: Drug: Lidocaine spray

INTERVENTIONS:
Drug: Lidocaine spray — Comparison of the success rate of endotracheal intubations between lidocaine spray and placebo
  Other Names: Placebo

SUMMARY:
This study aims to determine the first-pass success rate in video laryngoscopy and other parameters that topical anesthesia can affect during intubation.

DETAILED DESCRIPTION:
In Thailand, conventional intubation or sedation without paralysis is still the most common method of intubation due to the lack of emergency physicians at primary care centers. A pilot study had shown that topical oral anesthesia can improve the first-pass success rate in conventional intubation by direct laryngoscopy. This study aims to determine the first-pass success rate in video laryngoscopy and other parameters that topical anesthesia can affect during intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients in emergency department that have indication for conventional intubation
* Age > 18 yr

Exclusion Criteria:

* Patient who undergo RSI
* Patient who falls in cardiac arrest airway algorithm
* Patient who is currently pregnancy
* Known allergy to lidocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
First-pass success rate | 1 Year
  Comparison of the succession rate of endotracheal tube intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Savang Vadhana Memorial Hospital, Chon Buri, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: No